CLINICAL TRIAL: NCT03243552
Title: Proof of Mecahism Study for the Treatment of Social Anhedonia in ASD
Brief Title: Proof of Mechanism Study for the Treatment of Social Anhedonia in ASD
Acronym: ACEP4
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James McCracken, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACEPIV
Record Dates: First submitted 2017-07-27; First posted 2017-08-09 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: ASD

STUDY DESIGN:
Intervention Model Description: Phase IIa Proof of Mechanism 16-week, randomized, double-blind, controlled trial of L-DOPA versus placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L-DOPA versus Placebo (Active Comparator): L-DOPA or placebo (1:1 randomization). Dosing will begin at 25mg carbidopa/100mg L-DOPA in 3 divided doses, with a fixed-flexible titration schedule, allowing dose increases once per week of 100mg L-DOPA. Maximum dose is 600mg/d.
  Interventions: Drug: L-DOPA versus Placebo; Behavioral: Social Skills Training
- Social Skills (Experimental): All participants will receive 16-week manualized social skills training.
  Interventions: Drug: L-DOPA versus Placebo; Behavioral: Social Skills Training

INTERVENTIONS:
Drug: L-DOPA versus Placebo — Participants will be randomized in a blocked schedule to yield 1:1 L-DOPA: placebo assignment.
Behavioral: Social Skills Training — ASD participants will be enrolled concurrently in a 16-week manualized, structured, group-based, social skills training program (PEERS).
  Other Names: PEERS

SUMMARY:
This project will use the experimental medicine approach of a Phase IIa Proof of Mechanism 16-week, randomized, double-blind, controlled trial of L-DOPA versus placebo administration in combination with a 16 week social skills training group in order to: 1) identify differences in social reward processes in adolescent and young adult ASD participants versus healthy controls as measured by fMRI activation in reward circuitry; 2) provide evidence of dopaminergic moderating effects on social reward components in ASD with greater pre- to post-treatment changes expected in the subjects randomized to L-DOPA versus placebo; 3) examine the hypothesis that baseline readouts of putative dopamine signaling (wanting activation responses) will predict the extent of fMRI reward-related activation changes pre- to post-treatment; and, 4) examine the proposed relationship between pre- to post- L-DOPA fMRI reward changes and changes in individual self-report ratings of social wanting and ratings of videotaped positive affect in a structured interaction with an examiner. The study will enroll 56 participants with DSM-5 ASD between the ages of 13-30 years of age and 18 healthy control participants without histories of psychopathology for baseline comparisons.

DETAILED DESCRIPTION:
Participants will comprise two groups: 1) 56 (male and female) adolescents and young adults likely to meet inclusion/exclusion confirmed by study assessment who will be outpatients, ages 13 to 30 years, inclusive; and 2) 18 (male and female) healthy adolescents and young adults without any history of significant psychiatric disorders or treatment, who will be ambulatory, and will reflect the racial, ethnic, and socio-economic composition of Los Angeles, and will be recruited without regard to gender, race, or ethnic background.

Healthy control adolescents (and parents) and young adults who meet all inclusion and exclusion criteria, will undergo a one-day 4-5 hour research evaluation of current functioning and behavior, cognitive function, including intellectual testing, urine drug screen, completion of questionnaires about possible psychological symptoms, perform brief tests to measure reward response, and complete a research Magnetic Resonance Imaging scan. Healthy control will not receive any interventions or medication.

All eligible ASD participants will be enrolled concurrently in a 16-week, structured, group-based, social skills training program (PEERS®). After screening evaluations, eligible subjects will undergo baseline MRI scanning and behavioral assessments (self- and parent-report measures, videotaped interaction) and then randomized in a blocked schedule to yield 1:1 L-DOPA: placebo assignment, before beginning weekly social skills training. Medication administration will begin simultaneously with social skills training, and subjects will be seen weekly for the 1st 8 weeks, then biweekly for the final 4 weeks for safety assessments, dose titration, and compliance checks. During the 16-week study period, primary behavioral assessments will be repeated at Week 8 and at end of study on Week 16. A second MRI scan will be obtained within + 4 days of last social skills session. A follow-up safety phone call to assess post-study condition will be performed 30 days after completion of double-blind. The rich set of behavioral observations obtained across the 16 weeks will allow the possible identification of early clinical efficacy changes associated with L-DOPA administration, which could add further support for investigating this mechanism in future studies. Results from the project should inform reseacher's understanding of determinants of social dysfunction in ASD and may support further investigation of treatments modulating central nervous system dopamine function as a therapeutic strategy to enhance social functioning in ASD.

ELIGIBILITY:
Inclusion Criteria:

* ages 13 - 30 years inclusive;
* meets diagnostic criteria for ASD by clinical evaluation and ADOS;
* estimated FS IQ >70; 4) English reading ability of 6th grade;
* ability to participate and complete protocol expectations (fMRI scan, testing) in the examining clinician's judgment; and
* planned enrollment and acceptance for the UCLA PEERS® adolescent or young adult social skills training program.

Exclusion Criteria:

* significant perceptual deficits;
* need for continuation or anticipated of use of prohibited dopamine-modifying medications (stimulants, antipsychotics);
* presence of serious behavioral comorbidity such as aggression, major depressive disorder requiring additional intervention, or self-injurious behavior, or current of past history of suspected psychotic disorder;
* history of tic disorder;
* presence of significant medical illness which may impact CNS function.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in fMRI: Social Reward Task from Baseline to week 16 (4 months) | Baseline, week 16
  BOLD Activation: VS, ACC, OFC, Amygdala, Hippocampus (same units of measure)

SECONDARY OUTCOMES:
Change on Anticipatory and Consummatory Interpersonal Pleasure Scale Adolescent (ACIPS-A) | Baseline, week 8 (midpoint), week 16 (4 month/end of study)
  Total Score (change in score by timepoint; before treatment, midpoint, end)
Change on Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) | Baseline, week 8 (midpoint), week 16 (4 month/end of study)
  Total Score (change in score by timepoint; before treatment, midpoint, end)
Change on Child Behavior Checklist (CBCL) | Baseline, week 16 (4 month/end of study)
  T Scores of Syndrome Scales for ages 18 or under
Change on Youth Self Report (YSR) | Baseline, week 16 (4 month/end of study)
  T Scores of Syndrome Scales for ages 18 or under
Change on Adult Behavior Checklist (ABCL) | Baseline, week 16 (4 month/end of study)
  T Scores of Syndrome Scales for ages 18 or over
Change on SRS Self Report | Baseline, week 8 (midpoint), week 16 (4 month/end of study)
  Social Anhedonia
Change on SRS Parent Report | Baseline, week 8 (midpoint), week 16 (4 month/end of study)
  Social Anhedonia
change on Social Communication Interaction Test (SCIT) | Baseline, week 8 (midpoint), week 16 (4 month/end of study)
  6 subscales and total score (0-30)

CONTACTS AND LOCATIONS:
Overall Officials: James T McCracken, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No